CLINICAL TRIAL: NCT06889792
Title: A Proactive Approach to Prevent Non-communicable Diseases Through Screening and Educating Emergency Department Attendees to Adopt Healthy Lifestyles: A Randomised Clinical Trial
Brief Title: Prevent Non-communicable Diseases Through Screening and Educating Emergency Department Attendees to Adopt Healthy Lifestyles
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Li Ho Cheung William, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HMRF22230351
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Non Communicable Diseases; Health-risk Behaviours
Keywords: Health-risk Behaviours; Non Communicable Diseases; Emergency Department
MeSH Terms: conditions — Noncommunicable Diseases; Emergencies | interventions — Referral and Consultation; Models, Biological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WhatsApp/WeChat with video (Experimental): Participants in the intervention group will receive a brief health warning and advice on health-risk behaviours. In addition, they will be asked about their priority in engaging in healthy lifestyles. Moreover, participants will receive WhatsApp/WeChat messages during the first 6 months as a reminder to adhere to their desired healthy lifestyle and a link to a 1-minute video relevant to their selected healthy lifestyle.
  Interventions: Other: Theory of planned behaviour; Other: Foot-in-the-door technique; Other: Self-determination theory; Other: Follow-up booster intervention; Other: Practical Resource Hub for Healthy Life leaflet; Other: a brief intervention using the Ask, Warn, Advise, Refer and Do-it- again (AWARD) model
- Placebo (Placebo Comparator): Participants in the control group will receive brief advice on adopting healthy lifestyles through regular text messages.
  Interventions: Other: Practical Resource Hub for Healthy Life leaflet; Other: a brief intervention using the Ask, Warn, Advise, Refer and Do-it- again (AWARD) model

INTERVENTIONS:
Other: Theory of planned behaviour — This theory holds that an intention to engage in a health-related behaviour is determined by the proximal factors of attitudes, subjective norms, and perceived behavioural control. Attitudes represent individuals perceived likelihood of performing and appraisal of the consequences of performing a health-promoting behaviour. Subjective norms are the social pressure perceptions to either perform or not perform a health-promoting behaviour. Finally, perceived behavioural control is an individual's perception of control regarding performing the behaviour.
  Arms: WhatsApp/WeChat with video
Other: Foot-in-the-door technique — The foot-in-the-door technique, which was introduced by Freeman and Fraser, emphasises the notion that individuals who initially comply with a small, easy request are more likely to later comply with a larger request. Compliance with the first request or target increases the individual's confidence and alters their self-perceived capability and willingness regarding further requests or targets. This technique can facilitate the recruitment process and enhance compliance.
  Arms: WhatsApp/WeChat with video
Other: Self-determination theory — According to self-determination theory, behavioural regulation is more autonomous when it is internalised, as opposed to being regulated by external factors. Compared with external regulation, autonomous regulation is associated with increased self-efficacy, greater behavioural persistence, longer-term behavioural changes and more positive health behaviour. Autonomy is another influential determinant of behaviour that is emphasised by freedom of choice. There is some evidence that people who have greater autonomy demonstrating greater competence and self-efficacy in achieving behavioural change compared with those with less autonomy. As a result, increased autonomy will facilitate a gradual change in risky behaviours.
  Our intervention aims to first change the participants' attitudes and their subjective norms through risk communication. Using foot-in-the-door technique and self-determination theory, it will then increase participants' willingness to adopt a healthy lifestyle.
  Arms: WhatsApp/WeChat with video
Other: Follow-up booster intervention — Staff will send WhatsApp/WeChat messages approximately once a week to remind the participants to adhere to their desired health-related lifestyle for the first 6 months. In addition, during the first week, the RA will send participants a link via WhatsApp/WeChat to a 1-minute video developed by the research team comprising content relevant to their selected health-related lifestyle. Four separate 1-minute videos will be compiled, each focusing on a different healthy lifestyle. These videos will indicate the health hazards of continuing this health risk behaviour and the benefits of adopting a healthy lifestyle. Moreover, the RA will encourage the participants to watch the video and ask any questions regarding the video content via WhatsApp/WeChat.
  Arms: WhatsApp/WeChat with video
Other: Practical Resource Hub for Healthy Life leaflet — The participants will be provided a Practical Resource Hub for Healthy Life leaflet containing information on various applications, including (i) 'Move Your Body', (ii) 'Eat Healthy', (iii) 'Live Alcohol Free', and (iv) 'Stay Away from Tobacco', which were developed by the Hong Kong Department of Health
Other: a brief intervention using the Ask, Warn, Advise, Refer and Do-it- again (AWARD) model — The participants will receive a brief intervention using the Ask, Warn, Advise, Refer and Do-it- again (AWARD) model : (1) Ask about and assess health-risk behaviours; (2) Warn about the high morbidity and mortality risks associated with health-risk behaviours; (3) Advise on adopting healthy lifestyles to improve the participant's health; (4) Refer to hotline services, such as those for smoking cessation and alcohol treatment or the nearest district health centre to follow up their health status; and (5) Do it again if participants have not adopted a healthy lifestyle at follow-ups.

SUMMARY:
Objective: To examine the effectiveness of a general health promotion intervention based on self-determination theory in proactively helping emergency department (ED) attendees to adopt healthy lifestyles.

Hypothesis to be tested: A general health promotion intervention based on self-determination theory will be effective in helping people adopt healthy lifestyles.

Design and subjects: The investigators will conduct a randomised controlled trial involving 1,172 ED attendees from five major acute care hospitals in Hong Kong.

Instruments: A behavioural risk factor questionnaire will be used to identify participants' health risk behaviours and document their blood pressure and body mass index. The EuroQoL 5-Dimension 5-level will be used to assess participants' quality of life.

Interventions: Participants in the intervention group will receive a brief health warning and advice on health-risk behaviours. In addition, participants will be asked about their priority in engaging in healthy lifestyles. Moreover, participants will receive WhatsApp/WeChat messages during the first 6 months as a reminder to adhere to their desired healthy lifestyle and a link to a 1-minute video relevant to their selected healthy lifestyle. Participants in the control group will receive brief advice on adopting healthy lifestyles through regular text messages.

Main outcome measures: The number of healthy lifestyles adopted at 6 months. Data analysis and expected results: SPSS for Windows will be used for quantitative data analysis. A significantly higher proportion of participants in the intervention group will adopt healthy lifestyles and exhibit better quality of life than those in the control group at 6 and 12 months.

DETAILED DESCRIPTION:
Study design An assessor-blinded, multicentre RCT with a two-group between-subjects design will be used following the Consolidated Standards of Reporting Trial.

Setting The proposed project will be conducted at the EDs of five major acute care hospitals in different clusters in Hong Kong.

Recruitment At the EDs The investigators has obtained ethical approval from the institutional review boards of the five hospitals. All potential participants will be approached by emergency nurses before being discharged from the EDs. These nurses will provide potential participants with a leaflet detailing the nature, purpose, design, procedures, and potential benefits and risks of the study. Subsequently, the emergency nurses will refer the potential participants to the RA. Informed written consent will be obtained from all participants. Participants will be assured that their participation will be voluntary, with no prejudice attached to refusal, and that the information provided by them will be kept confidential. A baseline assessment will be performed using questionnaires. Then, participants will be informed that participants will receive a telephone call from an RA within 3 days to evaluate their potential health-risk behaviours and provide them with appropriate health advice to adopt healthy lifestyles. In addition, the participants will be provided a Practical Resource Hub for Healthy Life leaflet containing information on various applications, including (i) 'Move Your Body', (ii) 'Eat Healthy', (iii) 'Live Alcohol Free', and (iv) 'Stay Away from Tobacco', which were developed by the Hong Kong Department of Health

Intervention

1. Intervention group Brief intervention via telephone (within 3 days after visiting the ED) The participants will receive a brief intervention using the Ask, Warn, Advise, Refer and Do-it- again (AWARD) model, which was originally developed for primary-care tobacco cessation. This intervention includes the following steps: (1) Ask about and assess health-risk behaviours; (2) Warn about the high morbidity and mortality risks associated with health-risk behaviours; (3) Advise on adopting healthy lifestyles to improve the participant's health; (4) Refer to hotline services, such as those for smoking cessation and alcohol treatment or the nearest district health centre to follow up their health status; and (5) Do it again if participants have not adopted a healthy lifestyle at follow-ups. For the advice step, the RA will ask about the participants' priority in engaging in a desired health-related lifestyle based on their responses in the behavioural risk factor questionnaire. The participants will also be asked to choose a goal that the participants consider most attainable, such as quitting or reducing smoking, consuming more vegetables or less fatty foods or sugary drinks, performing more exercise, or reducing alcohol consumption. Although the participants will be encouraged to adopt aspects of a healthy lifestyle sequentially, the participants will have the option to adopt them simultaneously if the participants feel confident in doing so. Each participant will receive a brief (approximately 5 minutes) individual intervention providing health advice on their selected lifestyle goal. The entire intervention will last approximately 10 minutes and may be extended if necessary.

   At the end of the telephone call, the participant will be informed that the RA will assist them in achieving their health-related goals throughout the study by sending messages via

   WhatsApp/WeChat. Follow-up booster intervention (up to 6 months) During the first 6 months of the proposed project, the RA will send WhatsApp/WeChat messages approximately once a week to remind the participants to adhere to their desired health-related lifestyle. Instant messaging via mobile applications was found to be effective in enhancing treatment compliance. In addition, during the first week, the RA will send participants a link via WhatsApp/WeChat to a 1-minute video developed by the research team comprising content relevant to their selected health-related lifestyle. Four separate 1-minute videos will be compiled, each focusing on a different healthy lifestyle. These videos will indicate the health hazards of continuing this health risk behaviour and the benefits of adopting a healthy lifestyle. Moreover, the RA will encourage the participants to watch the video and ask any questions regarding the video content via WhatsApp/WeChat. One advantage of using videos to deliver instant health advice messages is the use of sound and images, which can elicit emotions, enhance understanding of abstract concepts, and improve the retention of new information through auditory, visual, and verbal stimulation. Moreover, the delivered content can be viewed by the participants at their convenience and own pace.

   Follow-up assessment of behavioural changes at 3, 6, and 12 months The success of the participants in achieving their targeted health-related lifestyle will be assessed through phone calls at 3, 6, and 12 months. If the participants report the successful adoption of a healthy lifestyle, the RA will encourage them to adopt another healthy lifestyle. Then, the RA will provide participants with brief healthcare advice (approximately 5 minutes) and send via WhatsApp/WeChat another 1-minute video focused on their newly chosen and desired health-related lifestyle.
2. Control group Participants will receive a brief telephone intervention based on the AWARD model from the trained RA, similar to that delivered to the intervention group. However, the RA will only advise the participants to adopt a healthy lifestyle. In addition, the RA will send regular SMS messages to participants at a frequency similar to that used for the intervention group. However, these messages will contain only general health advice. In addition, the participants will receive follow-up outcome assessments at the same schedule as that followed in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* being aged ≥18 years old Chinese
* being triaged as semi-urgent (level 4) or non-urgent (level 5) and discharged home on the same day after receiving medical attention
* having at least one health risk behaviour (tobacco use, harmful alcohol consumption, unhealthy diet, and physical inactivity)
* owning a smartphone and having an ability to use instant messaging applications (e.g. WhatsApp or WeChat).

Exclusion Criteria:

* having a poor cognitive state or mental illness
* being diagnosed with NCDs and undergoing regular follow-ups in outpatient clinics
* participating in another related study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1172 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
The composite event rate of adopting at least one of the four healthy lifestyles at 6 months. | from baseline to 6 months
  The composite event rate of adopting at least one of the four healthy lifestyles at 6 months which is measured by using a behavioural risk-factor questionnaire. The higher rate of adopting at least one of the four healthy lifestyles indicate the more successful to help emergency department attendees to adoption of a healthy lifestyle and lead healthier lives.

SECONDARY OUTCOMES:
The composite event rate of adopting at least one of the four healthy lifestyles adopted at 12 months | from baseline to 12 months
  The composite event rate of adopting at least one of the four healthy lifestyles adopted at 12 months which is measured by using a behavioural risk-factor questionnaire. The higher rate of adopting at least one of the four healthy lifestyles indicate the more successful to help emergency department attendees to adoption of a healthy lifestyle and lead healthier lives.
Improvement in health-related quality of life at 6 months | from Baseline to 6 months
  Participants' change of health-related quality of life between baseline and 6-month follow-ups will use EuroQol 5-level scale (EQ-5D-5L) to measure the quality of life. It consists of two part. The first part has 5 questions and each question has choices 1 to 5. Large number means a worse outcome in the first part. The second part has one question which is a scale of 0 to 100. Large number means a better outcome in the second part.
Improvement in health-related quality of life at 12 months | from baseline to 12 months
  Participants' change of health-related quality of life between baseline and 12-month follow-ups will use EuroQol 5-level scale (EQ-5D-5L) to measure the quality of life. It consists of two part. The first part has 5 questions and each question has choices 1 to 5. Large number means a worse outcome in the first part. The second part has one question which is a scale of 0 to 100. Large number means a better outcome in the second part.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, PhD, Principal Investigator — The Nethersole School of Nursing, CUHK
Locations (1):
- The Nethersole School of Nursing, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The relevant anonymized patient level data, full dataset, technical appendix, and statistical code are available on reasonable request. The approval from the Principal Investigator for the purpose of data use is required.
Time Frame: After the project has been completed and the results of the project has been published
Access Criteria: Request could be sent to Principal Investigator (williamli@cuhk.edu.hk)

REFERENCES:
- [Derived] Li WHC, Wong EL, Xia W, Chen H, Tsui SH, Chan YC, Cheung KY, Leung YF, Ho LKL, Choi KC, Chung OJ. A proactive approach to prevent non-communicable diseases through screening and educating emergency department attendees to adopt healthy lifestyles: Study protocol for a pragmatic, multicenter, randomized controlled trial. PLoS One. 2025 Jul 3;20(7):e0327558. doi: 10.1371/journal.pone.0327558. eCollection 2025. PMID 40608754